CLINICAL TRIAL: NCT06308757
Title: The Role of Very Low Calorie Ketogenic Diet (VLCKD) in Patients Affected by Non-Alcoholic Steatohepatitis (NASH) With Significant Fibrosis (KETONASH)
Brief Title: Role of the Very Low Calorie Ketogenic Diet (VLCKD) in Patients With Non-Alcoholic Steatohepatitis (NASH) With Fibrosis
Acronym: KETONASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Fabio Piscaglia, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 495/2021/Sper/AOUBo
Record Dates: First submitted 2024-02-19; First posted 2024-03-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: NASH; NAFLD; Obesity; Liver Fibrosis
Keywords: vlckd; diet; ketogenic diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Multicentric, Prospective, Open, Randomized, Controlled, and Interventional, with no medicinal use
Masking Description: Two-arms, 2: 1 randomization stratified by type 2 diabetes mellitus and gender
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLCKD arm (Experimental): The VLCKD dietary intervention consists of five phases:
  Ketogenic Low-Calorie Period (2 months):
  * Phase 1 (30 days - Visits 1-3): Ketogenic diet with low-fat content, 600 kcal/day.
  * Phase 2 (15 days - Visit 5): 660 kcal/day.
  * Phase 3 (15 days - Visit 5): 730 kcal/day
  Low-Calorie Period (2 months):
  Phase 4 (30 days - Visits 6-7): Hypocaloric diet with the reintroduction of different foods, 1,050 kcal/day.
  - Phase 5 (30 days - Visits 7-8): 1,400 kcal/day.
  During these phases, the patient will receive nutritional supplementation with vitamins, trace elements, and omega-3 fatty acids. Throughout the very low-calorie ketogenic period, the patient will have three interim dietetic consultations (Visits 2-4) and a medical visit (Visit 5). During the low-calorie period, the patient will receive alternating two dietetic consultations (Visits 6 and 7) and one medical visit every 30 days (Visit 8).
  Interventions: Dietary Supplement: Very-low-calorie ketogenic diet (VLCKD) with meal replacements
- Control LCD arm (Active Comparator): The control LCD arm consists of a diet with natural low-calorie foods (1200-1500 kcal/day or a reduction of 500-1000 kcal/day compared to baseline) and a low glycemic index based on the "Mediterranean Diet" model, following the most recent guidelines on MAFLD/NAFLD. Similar to the VLCKD arm, for the entire duration of the dietetic treatment, the patient will alternately receive dietetic consultations and medical visits.
  At the end of the dietary intervention, patients from both study arms will continue with a controlled, low glycemic index diet tailored to the patient's basal metabolic rate (BMR) (estimated with bioimpedance assessment) for an additional six months.
  Both study arms will follow a physical activity schedule and will have psychological-motivational support.
  Interventions: Dietary Supplement: Mediterranean low-calorie diet (LCD)

INTERVENTIONS:
Dietary Supplement: Very-low-calorie ketogenic diet (VLCKD) with meal replacements — The VLCKD study arm will receive an experimental diet therapy with very-low-calorie ketogenic meal replacements (VLCKD) consisting of 5 successive phases (600 - 1500 kcal/day).
  Arms: VLCKD arm
Dietary Supplement: Mediterranean low-calorie diet (LCD) — The Control arm LCD will receive standard Mediterranean type low-calorie diet (LCD) therapy by the most recent guidelines on MAFLD/NAFLD (1200-1500 kcal/day).
  Arms: Control LCD arm

SUMMARY:
The purpose of the KETONASH study is to evaluate, in patients with metabolic-associated fatty liver disease (MAFLD) with non-alcoholic steatohepatitis (NASH) and significant liver fibrosis, the effect of a very low-calorie ketogenic diet (VLCKD) compared to that of a standard low-calorie diet (standard Mediterranean LCD - in accordance with the European Association for the Study of the Liver/European Society for Clinical Nutrition and Metabolism guidelines on MAFLD/NAFLD).

DETAILED DESCRIPTION:
The KETONASH study is a multicenter, open-label, randomised, controlled clinical trial that will be consecutively proposed to all patients with histological diagnosis of non-alcoholic steatohepatitis (NASH) and significant hepatic fibrosis in the context of chronic metabolic liver disease (MAFLD/NAFLD).

Once the inclusion criteria are confirmed and the exclusion criteria are ruled out, patients will be subsequently randomly assigned (randomisation) with a 2:1 ratio to one of the two study arms:

* VLCKD Study Arm → will receive experimental diet therapy with very low-calorie ketogenic meals (VLCKD) consisting of 5 successive phases (600 - 1500 kcal/day).
* LCD Control Arm → will receive standard low-calorie diet therapy, a Mediterranean-type diet in accordance with the most recent guidelines on MAFLD/NAFLD (1200-1500 kcal/day).

The KETONASH study consists of an initial 4-month diet intervention phase (Visits 1-8), followed by a second 8-month weight maintenance phase (Visits 9-15). In both study arms, the intervention will be conducted through a standardised multidisciplinary approach (Physician/Dietitian/Nurse/Psychologist) aimed at weight loss through changes in dietary regimen, exercise program, and emotional support techniques.

The two study arms differ in nutritional composition, types of foods, and caloric intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with histological diagnosis of NASH with evidence of fibrosis (defined according to NASH CRN) obtained no more than 6 months before enrollment;
* Stable weight for more than 6 months with BMI between 30-40 kg/m2;
* Patients in whom it is safe and feasible to proceed with liver biopsy and who consent to undergo liver biopsy after 12 months of enrollment to assess the effect of dietary treatment;
* Obtained informed consent.

Exclusion Criteria:

* BMI <30 or BMI >40
* Presence of evolved chronic liver disease into cirrhosis (histological F4 or elastometric LSM >14 kPa)
* Type 1 diabetes mellitus
* Model for End-stage Liver Disease (MELD) score >12, AST or ALT ≥5× ULN, HbA1c >9.5%, INR ≥1.4, creatinine >1.5 mg/dl, platelets <100,000/mm3, and total bilirubin >1.5 mg/dl.
* Concurrent presence of any other known chronic liver disease beyond MAFLD/NAFLD, such as alcoholic liver disease, viral (HCV/HBV), cholestatic-autoimmune (PBC/PSC/AIH), Wilson's disease, hemochromatosis, drug-induced liver injury (DILI), or the presence or suspicion of hepatocellular carcinoma (HCC);
* Average alcohol consumption exceeding 4/2 units/day (males/females) in the preceding 6 months and a history of excessive alcohol consumption in the last 5 years;
* Previous or planned liver transplant, bariatric surgery, ileal resection, or biliary diversion;
* History of acute cholecystitis and biliary obstructions (cholangitis);
* Recent (in the last 12 months) or concurrent use of agents known to cause hepatic steatosis (long-term systemic corticosteroids [>10 days], amiodarone, methotrexate, tamoxifen, tetracyclines, high-dose estrogens, valproic acid);
* Recent (in the last 3 months) change in the dose/regimen or introduction of Vitamin E (at doses ≥400 IU/day), ursodeoxycholic acid (UDCA), betaine, S-adenosyl methionine, silymarin, or pentoxifylline;
* Presence of psychiatric disorders and/or diagnosis of any eating disorder;
* Life expectancy <6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Change of at least one grade of liver fibrosis | 12 months
  Histological change of liver fibrosis without worsening of NASH
Change of histological features of NASH | 12 months
  NASH parameters variation. Improvement in disease activity is defined as decrease in NAFLD Activity Score (NAS) ≥1 points. The worsening of fibrosis is defined as any numerical increase in the stage.

SECONDARY OUTCOMES:
Histological NIH NASH CRN Score | 12 months
  Assessment of individual histological components that make up the NIH NASH CRN (NASH Clinical Research Network) Score. NAS (NAFLD Activity Score) is the unweighted sum of steatosis, lobular inflammation, and hepatocellular ballooning scores. NAS of ≥5 correlated with a diagnosis of NASH, and biopsies with scores of less than 3 were diagnosed as not NASH.
Histological FLIP/SAF changes | 12 months
  Assessment of individual histological components that make up the FLIP (fatty liver inhibition of progression) SAF (steatosis activity fibrosis) score (based on steatosis, ballooning, lobular inflammation, fibrosis, etc.). The score ranges from 0 (not NAFLD) to 3 (NASH).
Biochemical test changes 1 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: aspartate transaminase (AST). Normal range: <50 U/L
Biochemical test changes 2 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: alanine aminotransferase (ALT). Normal range: <45 U/L
Biochemical test changes 3 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: Alkaline Phosphatase (range variable according to age and sex)
  Normal range:
  Females: 30 - 120 U/L Males: 30 - 120 U/L
Biochemical test changes 4 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: Gamma-glutamyltransferase
  Normal range:
  Females: < 38 U/L Males: < 55 U/L
Biochemical test changes 5 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: bilirubin Normal range: < 1.60 mg/dL
Biochemical test changes 6 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: glycemia (glucose) Normal range: 70 - 105 mg/dL
Biochemical test changes 7 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: HDL cholesterol
  Normal range:
  Females > 45 mg/dL Males > 35 mg/dL
Biochemical test changes 8 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: LDL cholesterol
  Normal range:
  Very high risk: objective < 55 high risk: < 70 moderate risk: < 100 low risk: < 116
Biochemical test changes 9 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: albumin Normal range: 35.0 - 50.0 g/L
Biochemical test changes 10 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: total proteins Normal range: 6.6 - 8.3 g/dL
Biochemical test changes 11 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: glicate hemoglobin Normal range: 20 - 42 mmol/mol
Biochemical test changes 12 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: Vitamin D Normal range: 15.2 - 90.1 pg/mL
Biochemical test changes 13 | 12 months
  Evaluation of variation of the biochemical tests panel based on normal ranges provided by the local laboratory. Multiple parameters are included in biochemical panel: uric acid
  Normal range:
  Females 2.4 - 5.7 Males 3.4 - 7.0 mg/dL
Fibrosis-4 test (FIB-4 ) variation | 12 months
  Liver biochemical biomarker (FIB4) variation
NAFLD Fibrosis Score (NFS) change | 12 months
  Liver biochemical biomarker (NAFLD Fibrosis Score, NFS) change
FAST (FibroScan-AST) score variation | 12 months
  Liver biochemical biomarker (FibroScan-AST) variation
Fatty Liver Index (FLI) modification | 12 months
  Liver biochemical biomarker (Fatty Liver Index (FLI) modification
Changes in LSM | 12 months
  Changes in physical liver biomarkers of fibrosis with Transient Elastometry (Fibroscan, Echosens, France) by reducing the kPa after treatment.
Variation of steatosis by CAP | 12 months
  Changes in biomarker of fatty liver disease evaluated with the controlled attenuation parameter (CAP, Echosens, France) by the reduction of decibel/sec (dB/sec) after treatment
Body Mass Index (BMI) improvement | 12 months
  Anthropometric parameters (BMI) improvement
Side effects evaluation for VLCKD therapy by VAS (Visual Analogue Scale) | 3 months
  The tolerability measured by a VAS (Visual Analogue Scale) that assesses the occurrence of side effects in patients undergoing diet therapy with VLCKD. The lowest value (0) indicates the best result, while the highest value (10) indicates absence of tolerability.
Compliance to VLCKD evaluated by VAS (Visual Analogue Scale) | 3 months
  The tolerability measured by a VAS (Visual Analogue Scale) that assesses the compliance of patients undergoing diet therapy with VLCKD. The lowest value (0) indicates the best result, while the highest value (10) indicates absence of tolerability.
Variation of steatosis by ultrasound assessment | 12 months
  Physical biomarkers of hepatic steatosis evaluated by qualitative method (mild, moderate, severe) hepatic ultrasound.
Questionnaires 1 | 12 months
  Questionnaires on quality of life (Health-related quality of life, HRQoL). The answers follow this scheme: 1 ["best outcome"] to 3 ["worst outcome"].
Questionnaires 2 | 12 months
  Questionnaires on lifestyle (physical exercise/sedentary habits). A score is not provided.
Questionnaires 3 | 12 months
  Questionnaires on liver disease-related events (NASH-CHECK). 0=no pain, 10=worst pain.
Questionnaires 4 | 12 months
  Questionnaires on liver disease-related events (CLDQ). 1=always, 7=never.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Piscaglia, Principal Investigator — University of Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT06308757/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT06308757/ICF_001.pdf